CLINICAL TRIAL: NCT01831817
Title: A Proof of Concept Study to Evaluate the Efficacy of an Occlusion Based Dentifrice in the Relief of Dentinal Hypersensitivity
Brief Title: Exploratory Study to Evaluate the Efficacy of an Occlusion Based Dentifrice in Relief of Dentinal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RH01591
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-02

CONDITIONS: Dentinal Hypersensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5% calcium sodium phosphosilicate/ sodium monofluorophosphate (Experimental): Dentifrice containing 5.0% w/w calcium sodium phosphosilicate and 1500ppmF as sodium monofluorophosphate
  Interventions: Drug: 5% calcium sodium phosphosilicate/ sodium monofluorophosphate dentifrice
- 0% calcium sodium phosphosilicate/sodium monofluorophosphate (Active Comparator): Dentifrice containing 0% w/w calcium sodium phosphosilicate and 1500ppmF as sodium monofluorophosphate
  Interventions: Drug: 0% calcium sodium phosphosilicate/ sodium monofluorophosphate dentifrice
- Sodium monofluorophosphate (Active Comparator): Dentifrice containing 1000 ppmF as sodium monofluorophosphate
  Interventions: Drug: Sodium monofluorophosphate dentifrice
- Sodium fluoride (Active Comparator): Dentifrice containing 1100 ppmF as sodium fluoride
  Interventions: Drug: Sodium Fluoride dentifrice

INTERVENTIONS:
Drug: 5% calcium sodium phosphosilicate/ sodium monofluorophosphate dentifrice — Calcium sodium phosphosilicate dentifrice (5% w/w) and 1500 ppm F as sodium monofluorophosphate
  Arms: 5% calcium sodium phosphosilicate/ sodium monofluorophosphate
Drug: 0% calcium sodium phosphosilicate/ sodium monofluorophosphate dentifrice — No calcium sodium phosphosilicate and 1500 ppm F as sodium monofluorophosphate
  Arms: 0% calcium sodium phosphosilicate/sodium monofluorophosphate
Drug: Sodium monofluorophosphate dentifrice — Sodium monofluorophospate dentifrice (1000 ppm F)
  Arms: Sodium monofluorophosphate
Drug: Sodium Fluoride dentifrice — Dentifrice containing 1100ppm F as sodium fluoride
  Arms: Sodium fluoride

SUMMARY:
The purpose of this exploratory study is to compare the treatment effect on dentinal hypersensitivity of a tubule occluding dentifrice as measured by Schiff and Tactile sensitivity. This proof of concept study will compare the test dentifrice with three other treatment groups.

DETAILED DESCRIPTION:
This will be a single center, eight week, randomized, controlled, examiner blind, four treatment arms, parallel design study in participants with at least two sensitive teeth that meet all the criteria at the Screening and Baseline visit. Participants will be assessed at baseline, four and eight weeks to monitor clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 55 years of age, in good general health, with pre-existing self-reported and clinically diagnosed tooth sensitivity are required for entry into the study.
* Participants will be required to have at least four teeth with facial/cervical erosion, abrasion and/or gingival recession which respond to qualifying evaporative (air) assessment at the Screening visit and have at least two teeth (incisors, canines or pre-molars) demonstrating signs of sensitivity, measured by qualifying tactile threshold (Yeaple ≤ 20 gram (g)) and evaporative (air) (Schiff Sensitivity Score ≥ 2) assessments at the Baseline visit.

Exclusion Criteria:

* Specific Dentition Exclusions for Test teeth

  1. Tooth with evidence of current or recent caries, or reported treatment of decay in 12 months of Screening.
  2. Tooth with exposed dentin but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing etiologies other than erosion, abrasion or recession of exposed dentin.
  3. Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator
* Use of a sensitivity dentifrice within 8 weeks of screening
* Individuals who require antibiotic prophylaxis for dental procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site
Pre-assignment Details: Participants aged 18 and 55 years of age (inclusive), in good general health, with preexisting self-reported and clinically diagnosed tooth sensitivity were enrolled in this study.
Groups:
- 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate: Dentifrice containing 5.0% w/w calcium sodium phosphosilicate and 1500ppm fluoride as sodium monofluorophosphate
- 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate: Dentifrice containing 0% w/w calcium sodium phosphosilicate and 1500ppm fluoride as sodium monofluorophosphate
- Sodium Monofluorophosphate: Dentifrice containing 1000 ppm fluoride as sodium monofluorophosphate
- Sodium Fluoride: Dentifrice containing 1100 ppm fluoride as sodium fluoride
Period: Overall Study
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Started | 35 | 34 | 35 | 36
Completed | 31 | 34 | 35 | 36
Not Completed | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawl of Consent | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT population consisted of all subjects who were randomized, administered at least one study treatment and provided at least one post-baseline assessment of efficacy. The data of 1 subject in 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate group who was lost to follow up was included in the ITT population.
Groups:
- 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate: Dentifrice containing 0% w/w calcium sodium phosphosilicate and 1500ppm fluoride as sodium monofluorophosphate
- Total: Total of all reporting groups
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride | Total
Number analyzed (Participants) | 32 | 34 | 35 | 36 | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (10.08) | 39.6 (9.72) | 38.3 (8.73) | 42.7 (9.10) | 39.5 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 28 | 30 | 118
  Male | 4 | 2 | 7 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Schiff Sensitivity Score at Week 4
Description: Response to a constant jet of air applied to hypersensitive teeth was evaluated using a Schiff Sensitivity pain response scale. According to this analog scale, pain response for each individual stimulated tooth ranged from 0 to 3; 0 - participant did not respond to air stimulation, 1 - participant responded to air stimulus but did not request discontinuation of stimulus, 2 - participant responded to air stimulus and requested discontinuation of stimulus, 3 - participant responded to air stimulus, considered stimulus to be painful and request discontinuation of stimulus.
Time Frame: Baseline and 4 weeks post administration of study treatment
Population: The ITT population was defined as all participants who were randomized, administered at least one study treatment during the study and had at least one post baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Number analyzed (Participants) | 32 | 34 | 35 | 36
Score on a scale
  Baseline | 2.39 (0.396) | 2.41 (0.435) | 2.40 (0.417) | 2.38 (0.403)
  Week 4 | 1.83 (0.779) | 1.94 (0.547) | 2.31 (0.516) | 2.31 (0.401)
  Mean change from baseline at Week 4 | -0.56 (0.759) | -0.47 (0.563) | -0.09 (0.445) | -0.07 (0.341)
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate; Principal null hypothesis to be tested was- H0: The change from baseline was the same for both treatments in all pairwise comparisons; Test type: Superiority or Other; p = 0.4321, ANCOVA; Mean change difference = -0.10, 95% CI 2-sided [-0.35 to 0.15] — Treatment as fixed factor and baseline Schiff score as covariate. Difference was First named treatment-second named treatment that a negative difference implied the mean of the second named treatment was larger than that of the first named treatment
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean change difference = -0.48, 95% CI 2-sided [-0.73 to -0.23] — Treatment as fixed factor and baseline Schiff score as covariate. Difference is First named treatment - second named treatment that a negative difference implies the mean of the second named treatment is larger than that of the first named treatment
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean change difference = -0.49, 95% CI 2-sided [-0.74 to -0.24] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Monofluorophosphate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0028, ANCOVA; Mean change difference = 0.38, 95% CI 2-sided [0.13 to 0.63] — Treatment as fixed factor and baseline Schiff score as covariate. Difference is second named treatment - first named treatment that a negative difference implies the mean of the first named treatment is larger than that of the second named treatment
Statistical Analysis 5: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Fluoride; Principal null hypothesis to be tested was- H0: The change from baseline waas the same for both treatments in all pairwise comparisons; Test type: Superiority or Other; p = 0.0022, ANCOVA; Mean change difference = 0.39, 95% CI 2-sided [0.14 to 0.63] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9606, ANCOVA; Mean change difference = -0.01, 95% CI 2-sided [-0.25 to 0.24] — [estimate comment as in outcome 1, analysis 4]

2. Primary Outcome: Mean Change From Baseline in Schiff Sensitivity Score at Week 8
Description: as for outcome 1
Time Frame: Baseline and 8 weeks post administration of study treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Number analyzed (Participants) | 32 | 34 | 35 | 36
Score on a Scale
  Baseline | 2.40 (0.396) | 2.41 (0.435) | 2.40 (0.417) | 2.38 (0.403)
  Week 8 | 1.60 (0.987) | 1.56 (0.894) | 2.41 (0.462) | 2.44 (0.427)
  Mean change from baseline at Week 8 | -0.81 (0.972) | -0.85 (0.901) | 0.01 (0.353) | 0.07 (0.450)
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8030, ANCOVA; Mean change difference = 0.04, 95% CI 2-sided [-0.30 to 0.38] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean change difference = -0.82, 95% CI 2-sided [-1.16 to -0.48] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean change difference = -0.86, 95% CI 2-sided [-1.20 to -0.53] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Monofluorophosphate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean change difference = 0.86, 95% CI 2-sided [0.53 to 1.19] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Fluoride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean change difference = 0.91, 95% CI 2-sided [0.58 to 1.23] — Treatment as fixed factor and baseline Schiff score as covariate. Difference is Second named treatment - first named treatment that a negative difference implies the mean of the second named treatment is larger than that of the first named treatment
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7872, ANCOVA; Mean change difference = -0.04, 95% CI 2-sided [-0.37 to 0.28] — [estimate comment as in outcome 1, analysis 4]

3. Primary Outcome: Median Change From Baseline in Tactile Sensitivity at Week 4
Description: Response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force was reached. The tactile threshold for each tooth was determined by asking the subject whether the sensation caused discomfort. The pressure setting at which the subject gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g.
Time Frame: Baseline and 4 weeks post administration of study treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: grams
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Number analyzed (Participants) | 32 | 34 | 35 | 36
grams
  Baseline | 10.00 [10.0 to 10.0] | 10.00 [10.0 to 10.0] | 10.00 [10.0 to 15.0] | 10.00 [10.0 to 15.0]
  Week 4 | 10.00 [10.0 to 45.0] | 10.00 [10.0 to 50.0] | 10.00 [10.0 to 15.0] | 10.00 [10.0 to 35.0]
  Median change from baseline at Week 4 | 0.00 [0.0 to 35.0] | 0.00 [0.0 to 40.0] | 0.00 [-5.0 to 5.0] | 0.00 [-5.0 to 20.0]
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.9642, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 0.00, 95% CI 2-sided [0.00 to 0.00] — Positive values favour the first named treatment
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.0016, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 0.00, 95% CI 2-sided [0.00 to 5.00] — Positive values favour the first named treatment
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.0100, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 0.00, 95% CI 2-sided [0.00 to 5.00] — Positive values favour the first named treatment
Statistical Analysis 4: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.0020, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 0.00, 95% CI 2-sided [0.00 to 0.00] — Positive values favour the second named treatment
Statistical Analysis 5: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.0122, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 0.00, 95% CI 2-sided [0.00 to 0.00] — Positive values favour the second named treatment
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.7138, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 0.00, 95% CI 2-sided [0.00 to 0.00] — Positive values favour the first named treatment

4. Primary Outcome: Median Change From Baseline in Tactile Sensitivity at Week 8
Description: as for outcome 3
Time Frame: Baseline and 8 weeks post administration of study treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: grams
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Number analyzed (Participants) | 32 | 34 | 35 | 36
grams
  Baseline | 10.00 [10.0 to 10.0] | 10.00 [10.0 to 10.0] | 10.00 [10.0 to 15.0] | 10.00 [10.0 to 15.0]
  Week 8 | 15.00 [10.0 to 90.0] | 15.00 [10.0 to 75.0] | 10.00 [10.0 to 55.0] | 10.00 [10.0 to 35.0]
  Median change from baseline at Week 8 | 5.00 [0.0 to 80.0] | 5.00 [0.0 to 65.0] | 0.00 [-5.0 to 45.0] | 0.00 [0.0 to 20.0]
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.9834, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 0.00, 95% CI 2-sided [-5.00 to 5.00] — Positive values favour the first named treatment
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.0001, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 5.00, 95% CI 2-sided [0.00 to 15.00] — Positive values favour the first named treatment
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.0003, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 2.50, 95% CI 2-sided [0.00 to 15.00] — Positive values favour the first named treatment
Statistical Analysis 4: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Test type: Superiority or Other; p < 0.0001, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = -5.00, 95% CI 2-sided [-10.00 to 0.00] — Positive values favour the second named treatment
Statistical Analysis 5: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.0002, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = -5.00, 95% CI 2-sided [-10.00 to 0.00] — Positive values favour the second named treatment
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.2894, Hodges-Lehmann Wilcoxon non-parametric; Hodges-Lehmann shift = 0.00, 95% CI 2-sided [0.00 to 0.00] — Positive values favour the first named treatment

5. Primary Outcome: Mean Change From Baseline in Visual Rating Scale Score at Week 4
Description: The intensity of response to stimulus will be rated using a 10 point scale where 1 denotes "No Pain" and 10 denotes "Intense Pain".
Time Frame: Baseline and 4 weeks post administration of study treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Number analyzed (Participants) | 32 | 34 | 35 | 36
Score on a scale
  Baseline | 6.66 (1.886) | 6.69 (1.723) | 6.41 (1.776) | 6.92 (1.783)
  Week 4 | 5.45 (2.212) | 5.72 (1.776) | 5.39 (1.702) | 6.38 (1.814)
  Mean change from baseline at Week 4 | -1.20 (1.727) | -0.97 (2.371) | -1.03 (1.356) | -0.54 (1.742)
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.5555, ANCOVA; Mean change difference = -0.24, 95% CI 2-sided [-1.03 to 0.56] — Treatment as fixed factor. Baseline Schiff strata and VRS as covariates. Difference is 1st named treatment - 2nd named treatment that a negative difference implies the mean of the 2nd named treatment is larger than that of the 1st named treatment
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.8769, ANCOVA; Mean change difference = -0.06, 95% CI 2-sided [-0.86 to 0.73] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.0562, ANCOVA; Mean change difference = -0.76, 95% CI 2-sided [-1.55 to 0.02] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.6562, ANCOVA; Mean change difference = -0.18, 95% CI 2-sided [-0.95 to 0.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.1788, ANCOVA; Mean change difference = 0.53, 95% CI 2-sided [-0.24 to 1.30] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.0734, ANCOVA; Mean change difference = -0.70, 95% CI 2-sided [-1.47 to 0.07] — [estimate comment as in outcome 5, analysis 1]

6. Primary Outcome: Mean Change From Baseline in Visual Rating Scale Score at Week 8
Description: as for outcome 5
Time Frame: Baseline and 8 weeks post administration of study treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Number analyzed (Participants) | 32 | 34 | 35 | 36
Score on a scale
  Baseline | 6.71 (1.892) | 6.69 (1.723) | 6.41 (1.776) | 6.92 (1.783)
  Week 8 | 4.65 (2.550) | 4.46 (2.076) | 5.70 (1.914) | 6.07 (2.046)
  Mean change from baseline at Week 8 | -2.06 (2.205) | -2.24 (2.287) | -0.71 (1.559) | -0.86 (1.673)
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.6727, ANCOVA; Mean change difference = 0.19, 95% CI 2-sided [-0.71 to 1.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.0072, ANCOVA; Mean change difference = -1.24, 95% CI 2-sided [-2.14 to -0.34] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.0056, ANCOVA; Mean change difference = -1.27, 95% CI 2-sided [-2.16 to -0.38] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Test type: Superiority or Other; p = 0.0016, ANCOVA; Mean change diference = 1.43, 95% CI 2-sided [0.56 to 2.31] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.0011, ANCOVA; Mean change difference = 1.46, 95% CI 2-sided [0.59 to 2.33] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Test type: Superiority or Other; p = 0.9413, ANCOVA; Mean change difference = -0.03, 95% CI 2-sided [-0.90 to 0.84] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Mean Change From Baseline in Dentine Hypersensitivity Experience Questionnaire Total Score at Week 4
Description: DHEQ Total score is an overall summary measure for the impact of dentine hypersensitivity on everyday life. Total score is calculated as the sum of 34 questions (each with a possible score of 1 to 7). The scale of responses range from 34 to 238. Higher values imply a worse outcome i.e. an increase in impact on dentine hypersensitivity on everyday life. Lower values imply a better outcome i.e. a decrease in impact on dentine hypersensitivity on everyday life.
Time Frame: Baseline and 4 weeks post administration of study treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Number analyzed (Participants) | 32 | 34 | 35 | 36
Score on a scale
  Baseline | 136.53 (34.194) | 132.55 (35.646) | 121.09 (44.467) | 133.89 (33.638)
  Mean change from baseline at Week 4 | -3.91 (21.850) | -4.39 (27.155) | -3.80 (24.874) | -7.50 (28.905)

8. Secondary Outcome: Mean Change From Baseline in Dentine Hypersensitivity Experience Questionnaire (DHEQ) Total Score at Week 8
Description: as for outcome 7
Time Frame: Baseline and 8 weeks post administration of study treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Number analyzed (Participants) | 32 | 34 | 35 | 36
Score on a scale
  Baseline | 134.33 (33.778) | 132.55 (35.646) | 120.09 (44.614) | 133.89 (33.638)
  Change from baseline at Week 8 | -6.43 (28.693) | -7.97 (31.324) | -3.88 (22.222) | -10.86 (33.669)

ADVERSE EVENTS:
Groups:
- 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate: DDentifrice containing 5.0% w/w calcium sodium phosphosilicate and 1500ppm fluoride as sodium monofluorophosphate
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34 | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 5/35 | 3/34 | 2/35 | 2/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate (N=35) | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate (N=34) | Sodium Monofluorophosphate (N=35) | Sodium Fluoride (N=36)
Headache (Nervous system disorders) | 1 (2) | 2 (2) | 1 (1) | 2 (2)
Arthralgia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in Jaw (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.